CLINICAL TRIAL: NCT07407868
Title: Evaluating The Impact on 90-day Survival Of Post-Discharge Follow-up Strategies Delivered To Adult Patients Hospitalized With Sepsis Across A Research Network In Sub-Saharan Africa
Brief Title: Call for Life Sepsis
Acronym: C4L-Sepsis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IDI-REC-2025-204
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Sepsis
Keywords: Reduce post discharge sepsis mortality,; Interactive Voice Response System,; Call for life - IVR
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Discharge Intervention (EDI) (No Intervention): 1. A standardized form provided around the time of hospital discharge (within 24 hours) with detailed information including the clinical course during hospitalization, including description of management and laboratory and clinical findings, discharge diagnosis, and any recommendations and treatment at discharge. The form will include a recommendation for a scheduled follow-up visit with a non-study clinician at the health facility from which the participant was discharged within 14 days after hospital discharge.
  2. Standardized information education communication (IEC) materials that include explanations and descriptions (e.g., pictorial depictions) of emergency signs for sepsis and key triggers for seeking care
- EDI plus IVR tool ( EDI-CFL IVR) (Experimental): EDI at the time of discharge, plus IVR tool: Participants will be provided analog phones with loaded airtime pro-rated to 3 months and instructions on battery charging. Features will include:
  1. Automated IVR using Call for Life for status checks and optional health information tips at day 0, 1, 2, 7 and every 7 days within the first 28 days, followed by every 14 days from day 29 to day 90.
  2. Reminders at 24 hours (day 13) and 48 hours (day 12) prior to scheduled appointments.
  3. Alerts mapped onto the dash board, the alerts may be due to missed clinic visit or symptoms reported by clients/participants. In case of a missed clinic, alert, the study clinician will inform the clinician in charge of client management to make a follow-up on the client who has missed a visit. In case of a symptom alert or report of symptoms requiring rapid follow-up, the study clinician gives medical advice to patients accordingly and this is documented in the system.
  Interventions: Other: Interactive Voice Response system-Call for life IVR

INTERVENTIONS:
Other: Interactive Voice Response system-Call for life IVR — The CFL-Sepsis system will be developed for this trial to provide sepsis-related health information tips for adult patients who have recovered from a sepsis hospitalization.
  In this trial, the IVR will be used to reach out to the participants through a phone call. The purpose of the IVR will be to help the patient report on any symptoms that will need a clinician's advice, the system will help deliver status checks on participants' well-being and deliver general information and health education on sepsis, including danger signs.
  Arms: EDI plus IVR tool ( EDI-CFL IVR)

SUMMARY:
Sepsis is a life-threatening organ dysfunction caused by a dysregulated host response to infection. Sepsis-attributable mortality in sub-Saharan Africa (sSA) is high, with in-hospital mortality in some settings approaching 40%. Studies show that mortality among children under 5 years hospitalized with sepsis remains high within the first 6 months of discharge. Additionally, high mortality has been observed among other populations within sSA, with factors such as HIV infection being associated with increased risk. Reducing sepsis deaths contributes to the achievement of the Sustainable Development Goals (SDG), particularly SDG 3 in reducing maternal mortality (3.1), neonatal and under five mortality (3.2), and burden of mortality from communicable diseases (3.3) and improving universal health coverage (3.8). The World Health Organization (WHO) has recognized sepsis as a global priority, with low- and middle-income settings being particularly affected. In sSA, sepsis is commonly associated with infectious diseases like malaria, Human Immunodeficiency Virus/ Acquired Immunodeficiency Syndrome (HIV/AIDS), pneumonia, tuberculosis, and diarrhea. Guidelines from the Surviving Sepsis Campaign (SSC) have become standard in some settings. However, little is known about patients' status post-discharge. This study aims to evaluate two post-discharge follow-up strategies for adult sepsis patients. Study duration is 45 months, participants will receive intervention up to 90 days post discharge.

Description of intervention: Post-discharge follow-up strategy 1: Enhanced Discharge Intervention (EDI) Post-discharge follow-up strategy 2: EDI plus Interactive Voice Response (IVR)

Objectives:

The study aims to evaluate two post-discharge follow-up strategies for adult patients hospitalized with sepsis, focusing on their efficacy in reducing the 90-day mortality, and their effect on return to follow-up, number of re-admissions, and quality of life.

Primary efficacy endpoint

* 90- day all-cause mortality post discharge Secondary end points
* Time to death
* 28-day all-cause mortality
* Attendance within 14-day check-up post discharge
* Re-admission within 28 and 90 days
* Days alive and out of hospital (DAOH)
* Quality of life score (Baseline vs 28 day and Baseline vs 90 days)
* Differences in baseline demographic and clinical characteristics (e.g., age, sex, disease severity, comorbidities, key laboratory values) between randomized participants and screen failures. Study design: This is an open-label, randomized, parallel, interventional study, with two post-discharge follow-up strategies: 1) EDI; or 2) EDI plus IVR system. Fixed allocation randomization at a 1:1 ratio will be applied to either study arm.

Sample size: A total of 1,410 (705 per arm) from the four countries (Uganda, Nigeria, Ghana and Mozambique) will be enrolled competitively across the sites.

ELIGIBILITY:
Inclusion Criteria:

* At admission

  1. Adults ≥18 years.
  2. Participant's hospital admission diagnosis is consistent with the following broad definition of sepsis, incorporating its principal components (signs of infection plus signs of severity/organ dysfunction):

     1. Signs of infection: Suspected or proven infection, as determined by the medical team in charge.
     2. Illness severity: Decision of the medical team to admit the patient to an adult medical ward of the study hospital, according to clinical appraisal of the treating physician and applicable guidelines.
  3. Participant/proxy is willing to have their medical records reviewed by the trial team and get daily follow-ups until the time of discharge and to be approached again by the study team for a second informed consent process towards the time of hospital discharge.
  4. Evidence of a personally signed and dated informed consent form stating that the participant/proxy has been informed of, had opportunity to ask questions about and have consented to the initial study procedures that will be conducted during their hospitalization. At discharge
  5. Patient has overcome the critically ill phase of their hospitalization and is, according to the non-study clinical team caring for the patient, expected to be discharged within the next 24 hours.
  6. Participant is willing and able to comply with scheduled phone follow-ups, and other study procedures.
  7. Evidence of a personally signed and dated informed consent form stating that the participant has been informed of, had opportunity to ask questions about and have consented to all procedures that will be conducted at the time of and after their discharge, and alternatives and risks for the study.
  8. The participant confirms that there is availability of mobile network coverage in their place of residence.

Exclusion Criteria:

At Admission;

1. Patient who requires hospitalization for a condition that requires emergent or urgent obstetric or surgical intervention (including burns, trauma, abscess)
2. Persons who are currently or have been previously enrolled into this study.
3. Patient is terminally ill due to an underlying condition other than sepsis.
4. The patient is a detainee or prisoner.
5. The patient is unable to speak English and Luganda.

   * At Discharge:

   At discharge
6. The patient is unable to hear.
7. Participant states they will be unable to return to same health facility for the scheduled 14-day post-discharge clinic assessment (provided by the non-study clinical team)
8. Patients requiring clinical care for more than 10 days (if clinical care was completed and participant is ready for discharge but are still in hospital for financial or logistical reasons beyond 10 days, they can still be eligible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1410 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2028-03-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality by Day 90 post-discharge (binary; time-to-event) | Day 90 post discharge
  To determine the effect of EDI + IVR versus EDI alone on 90-day all-cause mortality after hospital discharge

IPD SHARING:
Plan to Share IPD: Undecided
This needs teh TMG to decide and approval of Data sharing agreement by the Uganda National Council of Science and Technology